CLINICAL TRIAL: NCT02202148
Title: Liver Stiffness Measurement in Alcohol-dependent Subjects in Relation to Abstinence After Withdrawal
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Collaborators: Hôpital Dupuytren (Other)
Responsible Party: Principal Investigator, Philippe Nubukpo, MD, PhD, Centre Hospitalier Esquirol
Other Study IDs: 2014-A00854-43
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Alcohol Withdrawal
Keywords: Fibroscan; alcohol dependence; alcohol withdrawal; controlled attenuation parameter; BDNF
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- alcohol withdrawal

SUMMARY:
This study is complementary to the main study "Brain Derived Neurotrophic Factor Serum Levels Evolution During the Six Months After Alcohol Withdrawal " NCT01491347.

Liver stiffness variation is one of the major somatic effect of chronic alcohol consumption. It is a consequence of numerous mechanisms, including inflammation. Liver stiffness seems to depend on alcohol consumption in alcohol dependent patient, more precisely on the time after the last alcohol consumption. This is very few documented after alcohol withdrawal, and has never been explored during several months after withdrawal as a function of alcohol consumption and abstinence.

Brain Derived neurotrophic Factor (BDNF) seems to play a major role in general homeostasis and also liver function.

We propose here to analyse the serum BDNF levels variations after withdrawal according to liver stiffness levels and alcohol consumption status.

We will also measure liver stiffness using Fibroscan® in alcohol dependent subjects included in the main study to search for a link with serum BDNF levels and abstinence at day 0, 14, 28 and months 2, 4, and 6.

ELIGIBILITY:
Inclusion Criteria:

* participation to the study "BDNF serum levels evolution during 6 months after alcohol withdrawal" (main study)
* criteria from the main study

Exclusion Criteria:

* criteria from the main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: alcohol-dependent subjects hospitalized for alcohol withdrawal
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
BDNF serum levels as a function of stiffness categories in the abstinent and non abstinent groups at inclusion and at the different follow-ups of the study (M2, M4, M6) | 6 months maximum

SECONDARY OUTCOMES:
serum BDNF levels variations between inclusion and M2, M2 and M4 and M4 and M6. | 6 months
liver stiffness categories according to stiffness measurements at inclusion, M2, M4 and M6 | 6 months
Variations in liver stiffness | 6 months
controlled attenuation parameter (CAP) at each follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nubukpo, MD, PhD, Principal Investigator — Centre Hospitalier Esquirol
Locations (1):
- Centre Hospitalier Esquirol, Limoges, France